CLINICAL TRIAL: NCT05604586
Title: Assessment of the Impact of N-acetylcysteine Supplementation on Physical Performance Depending on the Polymorphism of Genes Related to Folate Metabolism
Brief Title: Assessment of the Impact of N-acetylcysteine Supplementation on Physical Performance
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Poznan University of Life Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: NAC/29112021
Record Dates: First submitted 2022-07-07; First posted 2022-11-03 (Actual); Last update posted 2022-11-03 (Actual); Status verified 2022-11

CONDITIONS: Skeletal Muscle Performance; Gene Polymorphisms
Keywords: Sport performance; gene polymorphism; N-acetylcysteine
MeSH Terms: interventions — Acetylcysteine

STUDY DESIGN:
Intervention Model Description: Eligible volunteers will be randomly assigned to one of the research groups. One of the groups will be taking the supplement for a period of 7 days, while the other group will be taking a placebo. Then a 3 week washout period will be performed. After that the groups will be exchanged and each participant will be assigned to a different group than it was in the first period of the study.
Who Masked: Participant, Investigator
Masking Description: Double (Participant/investigator)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- N-acetylcysteine (Experimental): Intervention: Dietary Supplement: N-acetylcysteine Participants will undergo two exercise tests and daily supplementation with N-acetylcysteine orally in three doses a day for seven consecutive days.
  Interventions: Dietary Supplement: N-acetylcysteine
- Placebo (Placebo Comparator): Supplement: Placebo Participants will undergo two exercise tests and daily supplementation with placebo orally in three doses a day for seven consecutive days.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: N-acetylcysteine — 100 women and men supplementing 1200 mg of N-acetylcysteine daily in three equal doses. Supplementation will last for 7 days.
  Arms: N-acetylcysteine
Dietary Supplement: Placebo — 100 women and men supplementing 1200 mg of placebo daily in three equal doses. Supplementation will last for 7 days.
  Arms: Placebo

SUMMARY:
Study aims to verify the hypothesis:

* N-acetylcysteine (NAC) supplementation improves exercise capacity in people training endurance sports and the effectiveness of this supplementation depends on the polymorphism of genes related to folate and glutathione metabolism.
* NAC supplementation affects the parameters of oxidative stress among women and men training endurance disciplines

DETAILED DESCRIPTION:
* Glutathione depletion caused by a combination of intense physical exertion associated with the generation of significant amounts of reactive oxygen species (ROS), and possibly with having an unfavorable variant of the methylenetetrahydrofolate reductase (MTHFR), glutamate-cysteine ligase catalytic subunit (GCLC); glutamate-cysteine ligase modifier subunit (GCLM); glutathione S-transferase Pi 1 (GSTP1); glutathione synthetase (GSS) or cystathionine-β-synthase (CBS) genes may contribute to lower adaptation to exercise, but also to deterioration of health of people training endurance sports.
* The main objective of the study is to verify the hypothesis that NAC supplementation has a beneficial effect on regeneration between intense exercise tests simulating a race characteristic for a given discipline. In addition, this study is aimed at checking whether genotype may modify the effectiveness of the supplementation measured as exercise and biochemical parameters . A double-blind study involving 100 women and men supplementing 1200 mg of N-acetylcysteine daily or 1200 mg of maltodextrin in three equal doses. Supplementation will last for 7 days. Blood sampling and body composition testing will be performed in the morning of the exercise test day. Discipline-specific exercise testing will be performed before and after the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Consent to participate in the study and acceptance of the established scheme for conducting the intervention
* age range between 18 and 45 years old
* regular training with a frequency of at least 4 times a week during the last year,

Exclusion Criteria:

* no consent to participate in the study and no acceptance of the established scheme of the conducted intervention
* existing diseases of the blood system and neoplastic diseases
* respiratory system diseases
* obesity
* any medical contraindications to exercise
* Results obtained from exercise tests that do not meet the inclusion criteria
* use of NAC during the last month
* allergy to NAC
* smoking
* pregnancy and lactation

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-05-01 (Actual); Primary Completion 2025-03-15 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Assesment of change in results of time trial test | Baseline,1 week
  (min/test) change within groups and between groups

SECONDARY OUTCOMES:
Reduced glutathione (GSH) | Baseline,1 week
  GSH (µM) concentrations change within the group and between the groups
Oxidized glutathione (GSSG) | Baseline,1 week
  GSSG (µM) concentrations change within the group and between the groups
Homocysteine (Hcy) | Baseline,1 week
  Hcy (µmol/l) concentrations change within the group and between the groups
Total cholesterol (TChol) | Baseline,1 week
  TChol (mg/dl) concentrations change within the group and between the groups
Blood HDL-cholesterol (HDL-C) | Baseline,1 week
  HDL-C (mg/dl) concentrations change within the group and between the groups
Blood LDL-cholesterol (LDL-C) | 1 week
  LDL-C (mg/dl) concentrations change within the group and between the groups
Blood triacylglycerol (TAG) | Baseline,1 week
  TAG (mg/dl) concentrations change within the group and between the groups
Dietary intake | Baseline,1 week
  macro and micronutrient intake (g,mg,ug)
aspartate aminotransferase (ASPAT) | 1 week
  ASPAT [U/l] Changes within groups and between groups
Alanine transaminase (ALAT) | Baseline,1 week
  ALAT [U/l] change within groups and between groups
Oxygen volume (VO2) | Baseline,1 week
  VO2 (ml/kg bw./min) change within groups and between groups
Carbon dioxide volume (VCO2) | Baseline,1 week
  VCO2 (ml/kgm.c./min) change within groups and between groups
Testosterone (T) | Baseline,1 week
  T (ng/dL) concentrations change within the group and between the groups
Cortisol (C) | Baseline,1 week
  C (ng/dL) concentrations change within the group and between the groups
Body mass(BM) | Baseline, 1 week
  Change in BM (kg) within groups and between groups
Fat Free Mass (FFM) | Baseline, 1 week
  FFM change within (kg) groups and between groups
Fat Mass% (FM%) | Baseline, 1 week
  FM% change within groups and between groups
Thiobarbituric Acid Reactive Species (TBARS) | 1 week
  TBARS concentrations change within the group and between the groups

CONTACTS AND LOCATIONS:
Overall Officials: Marcin Sadowski, MSc, Principal Investigator — Poznań University of Life Science
Locations (1):
- Poznan University of Life Science, Poznan, Poland

IPD SHARING:
Plan to Share IPD: No